CLINICAL TRIAL: NCT00896233
Title: Test-Retest Repeatability Study of Magnetic Resonance Elastography (MRE) for Liver Fibrosis Assessment in Healthy Volunteers and Hepatitis C Virus-Infected Patients
Brief Title: Magnetic Resonance Elastography for Assessment of Liver Fibrosis (MK-0000-132)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-132; 2009_588
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Liver Fibrosis; Hepatitis C Virus
Keywords: Staging of liver fibrosis prior to clinical trials for treatment of Hepatitis C Virus
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRE (Experimental)
  Interventions: Procedure: MRE

INTERVENTIONS:
Procedure: MRE — Part 1: Participants will have a screening visit, followed ~1 month later by two imaging visits over ~14 days. Each imaging visit will consist of two liver MRE scans.
  Part 2: Participants will have a screening visit, followed ~1
  month later by one imaging visit. The imaging visit will consist
  of two liver MRE scans.

SUMMARY:
This study will assess the repeatability of Magnetic Resonance Elastography (MRE) in both healthy volunteers and Hepatitis C Virus (HCV)-infected patients with fibrosis and lay the groundwork for the validation of MRE as an alternative to liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and at least 18 years of age
* Generally good health
* Willing to fast for 8 hours prior to each study visit

Hepatitis C Virus (HCV) Inclusion Criteria:

* Positive serology for HCV and detectable HCV ribonucleic acid (RNA) in blood within 12 weeks of screening;

For Part I, known fibrosis stage of at least =F2 (METAVIR) or =F3 (Ishak) from biopsy performed within 3 months of screening; For Part 2, known fibrosis stage of F1-F4 (METAVIR) or F1-F6 (Ishak)

* Never been treated for HCV

Healthy Participant Inclusion Criteria:

* Documented absence of hepatitis B virus, HCV, acute hepatitis A virus, and human immunodeficiency virus (HIV) within 12 weeks of screening

Exclusion Criteria:

* History of stroke, seizures, or neurological disorders
* Consumption of excessive amounts of alcohol
* Use of products containing nicotine
* Unable to hold a breath for 20 seconds
* Claustrophobia
* Use of illicit drugs or history of drug or alcohol abuse

HCV-Positive Exclusion Criteria:

* Evidence or history of chronic hepatitis not caused by HCV
* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Shire NJ, Yin M, Chen J, Railkar RA, Fox-Bosetti S, Johnson SM, Beals CR, Dardzinski BJ, Sanderson SO, Talwalkar JA, Ehman RL. Test-retest repeatability of MR elastography for noninvasive liver fibrosis assessment in hepatitis C. J Magn Reson Imaging. 2011 Oct;34(4):947-55. doi: 10.1002/jmri.22716. Epub 2011 Jul 12. PMID 21751289

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 2 of the study was not conducted; however, in Part 2 of the study, participants would have had a screening visit, followed ~1 month later by one imaging visit. The imaging visit would have consisted of two liver Magnetic Resonance Elastography (MRE) scans.
Groups:
- Magnetic Resonance Elastography (MRE): In Part 1 of the study, participants had a screening visit, followed ~1 month later by two imaging visits over ~14 days. Each imaging visit consisted of two liver MRE scans.
Period: Overall Study
Arm/Group | Magnetic Resonance Elastography (MRE)
Started | 10
Completed | 9
Not Completed | 1
Not completed — Claustrophobia during MRI | 1

BASELINE CHARACTERISTICS:
Arm/Group | Magnetic Resonance Elastography (MRE)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Repeated Maximum Liver Elastic Stiffness (Kilopascal [kPa]) Measurements
Description: Reader evaluated 4 sections of the liver at 4 different time points and the end result was a single region of interest (ROI) that could be measured in the registered elastograms at each of the time points. Stiffness measures obtained using the "Individual ROI" (average of the 4 individual ROI's selected by the reader, one for each slice of liver) and "Common ROI" (intersection (or area of common overlap) of the 4 individual ROI's) analysis methods were compared. The mean was the overall mean of the data and the standard deviation was the within participant standard deviation.
Time Frame: 14 days
Population: Participants analyzed were Completers.
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Reader 1: Participant scans evaluated by Reader 1.
- Reader 2: Participant scans evaluated by Reader 2.
Arm/Group | Reader 1 | Reader 2
Number analyzed (Participants) | 9 | 9
kPa
  MRE Common ROI | 4.54 (0.48) [0.82 to 0.99] | 4.64 (0.50) [0.72 to 0.98]
  MRE Individual ROI | 5.10 (0.44) [0.78 to 0.98] | 5.14 (0.41) [0.75 to 0.98]
Statistical Analysis 1: Comparison: Reader 1; ICC for measures of liver stiffness obtained by MRE (i.e., average over all 4 slices of the maximum stiffness for each slice) with respect to repeatability (precision) of multiple MRE assessments. This pertains to the Common ROI; Test type: Superiority or Other; ICC = 0.90, 90% CI 2-sided [0.81 to 0.99]
Statistical Analysis 2: Comparison: Reader 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ICC = 0.85, 90% CI 2-sided [0.71 to 0.98]
Statistical Analysis 3: Comparison: Reader 1; ICC for measures of liver stiffness obtained by MRE (i.e., average over all 4 slices of the maximum stiffness for each slice) with respect to repeatability (precision) of multiple MRE assessments. This pertains to the Individual ROI; Test type: Superiority or Other; ICC = 0.88, 90% CI 2-sided [0.78 to 0.98]
Statistical Analysis 4: Comparison: Reader 2; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ICC = 0.86, 90% CI 2-sided [0.75 to 0.98]

2. Primary Outcome: Repeated Mean Liver Elastic Stiffness (kPa) Measurements
Description: Reader evaluated 4 sections of the liver at 4 different time points and the end result was a single ROI that could be measured in the registered elastograms at each of the time points. Stiffness measures obtained using the "Individual ROI" (average of the 4 individual ROI's selected by the reader, one for each slice of liver) and "Common ROI" (intersection (or area of common overlap) of the 4 individual ROI's) analysis methods were compared. The mean was the overall mean of the data and the standard deviation was the within participant standard deviation.
Time Frame: 14 days
Population: Participants analyzed were Completers.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Reader 1 | Reader 2
Number analyzed (Participants) | 9 | 9
kPa
  MRE Common ROI | 3.12 (0.26) [0.80 to 0.99] | 3.14 (0.31) [0.78 to 0.99]
  MRE Individual ROI | 3.08 (0.19) [0.87 to 1.00] | 3.15 (0.20) [0.88 to 1.00]
Statistical Analysis 1: Comparison: Reader 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ICC = 0.90, 90% CI 2-sided [0.80 to 0.99]
Statistical Analysis 2: Comparison: Reader 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ICC = 0.88, 90% CI 2-sided [0.78 to 0.99]
Statistical Analysis 3: Comparison: Reader 1; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ICC = 0.93, 90% CI 2-sided [0.87 to 1.00]
Statistical Analysis 4: Comparison: Reader 2; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ICC = 0.94, 90% CI 2-sided [0.88 to 1.00]

3. Primary Outcome: Percent Difference in Mean Liver Stiffness Between Hepatitis C Virus (HCV)- Positive Participants With Liver Fibrosis and Healthy Participants
Description: Reader evaluated 4 sections of the liver at 4 different time points and the end result was a single region of interest (ROI) that could be measured in the registered elastograms at each of the time points. Stiffness measures obtained using the "Individual ROI" (average of the 4 individual ROI's selected by the reader, one for each slice of liver) and "Common ROI" (intersection (or area of common overlap) of the 4 individual ROI's) analysis methods were compared.
Time Frame: 14 days
Population: Participants analyzed were Completers.
Measure: Number (95% Confidence Interval); unit: percent treatment difference
Arm/Group | Reader 1 | Reader 2
Number analyzed (Participants) | 9 | 9
percent treatment difference
  MRE Common ROI | 94.41 [33.85 to 182.36] | 94.66 [32.65 to 185.67]
  MRE Individual ROI | 97.02 [39.77 to 177.73] | 99.31 [37.81 to 188.27]

4. Primary Outcome: Percent Difference in Maximum Liver Stiffness Between HCV- Positive Participants With Liver Fibrosis and Healthy Participants
Description: as for outcome 3
Time Frame: 14 days
Population: Participants analyzed were Completers.
Measure: Number (95% Confidence Interval); unit: percent treatment difference
Arm/Group | Reader 1 | Reader 2
Number analyzed (Participants) | 9 | 9
percent treatment difference
  MRE Common ROI | 117.21 [33.70 to 252.87] | 91.24 [32.12 to 176.83]
  MRE Individual ROI | 105.35 [38.51 to 204.42] | 90.77 [34.64 to 170.29]

ADVERSE EVENTS:
Arm/Group | Magnetic Resonance Elastography (MRE)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Resonance Elastography (MRE) (N=10)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Since both primary objectives were met based on the Part 1 analysis, a decision was made to stop the study and not proceed to Part 2. Therefore, data from Part 1 of the study were used for outcome measures 3 and 4 instead of data from Part 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications derived from this study should include input from the investigators and SPONSOR personnel.Such input should be reflected in publication authorship.The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts,or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.